CLINICAL TRIAL: NCT06084624
Title: Evaluation of Topical Rebamipide Versus Topical Betamethasone for Management of Oral Ulcers in Behcet's Disease: A Randomized Clinical Trial
Brief Title: Evaluation of Topical Rebamipide Versus Topical Betamethasone for Management of Oral Ulcers in Behcet's Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa Belal Omar Marzouk, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3623
Record Dates: First submitted 2023-10-10; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Oral Ulceration Due to Behçet's Disease
Keywords: Behcet Disease; Oral ulcers; oral ulceration
MeSH Terms: conditions — Behcet Syndrome; Oral Ulcer | interventions — rebamipide; Betamethasone

STUDY DESIGN:
Intervention Model Description: The study is a parallel 2 arm randomized controlled clinical trial where one group will be assigned to the rebamipide mouthwash, while the other group will be assigned to the betamethasone group randomly.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: the allocation of the participants to the groups will be concealed . The bottles of both mouthwashes will be the same. The solution of both mouthwashes will be of the same colour, odor and consistency.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rebamipide mouthwash (Experimental): Rebamipide mouthwash will be administered four times daily for one week or till healing
  Interventions: Drug: Rebamipide mouthwash
- Betamethasone mouthwash (Active Comparator): Betamethasone mouthwash of will be administered four times daily for one week or till healing
  Interventions: Drug: Betamethasone mouthwash

INTERVENTIONS:
Drug: Rebamipide mouthwash — Rebamipide (REB), 2-(4-chlorobenzoylamino)-3-[2(1H)-quinolinone-4-yl]-propionic acid, is commonly used in cases of gastric ulcers, gastritis, and dry eye syndrome
  Other Names: topical rebamipide
  Arms: Rebamipide mouthwash
Drug: Betamethasone mouthwash — Betamethasone is a potent glucocorticoid steroid. It is very soluble in water, and therefore it can be used as a mouthwash and has been used for symptomatic relief and treatment of recurrent aphthous ulcers
  Other Names: topical betamethasone
  Arms: Betamethasone mouthwash

SUMMARY:
The goal of this randomized clinical trial is to to compare the effect of topical rebamipide to topical betamethasone on oral ulcer severity in patients with Behcet's disease.. The main question it aims to answer is :

What is the effect of topical Rebamipide mouthwash compared to topical betamethasone mouthwash in management of oral ulcers in Behcet's disease?

Participants will will be divided randomly into the two groups and the following outcomes will be measured:

The oral ulcers severity Pain associated with oral ulcers Number of oral ulcers Healing time of oral ulcers

DETAILED DESCRIPTION:
This is a Randomized clinical trial (RCT) parallel groups, two arm, equivalence framework with 1:1 allocation ratio which is based on the hypothesis that Topical rebamipide has comparable effect to topical betamethasone on oral ulcer severity in patients with Behcet's disease The participants in this study will be recruited from the Rheumtology Clinic, Kasr el ainy hospital by HL as well as Oral Medicine Clinic and the dental Diagnostic center, Faculty of Dentistry, by MB. The eligible participants will be enrolled in the study in a consecutive order till the sample size is achieved.

Simple randomization will be generated using computerized random number generator (random.org) with allocation ratio (1:1).

Allocation concealment will be done using sequentially numbered opaque sealed opaque containers of the same shape, size and colour until interventions are assigned.

The entire procedure will be explained to the patients and a written consent will be obtained by the operator.

Participants and care givers will be blinded as both topical rebamipide and topical betamethasone mouthwashes will be of same consistency and will be provided in sealed opaque containers of the same shape, size and colour.

The enrolled patients will be divided randomly into two groups. One group will receive topical rebamipide mouthwash four times daily for one week or till healing and the other group will receive topical Corticosteroid (topical betamethasone) four times daily for one week or till healing. The patients will be recalled during the first week (days 1, 3, and 7), then every week for 3 weeks, afterward every month for 2 months. The patients will be asked to prohibit use of any topical medication during the trial. Outcome measures will be recorded in each visit.

Data will be analyzed using IBM SPSS advanced statistics (Statistical Package for Social Sciences), version 24 (SPSS Inc., Chicago, IL)

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with Behcet's disease as defined by the revised International Criteria for Behcet's Disease (ICBD2014).
2. Patients with active oral ulcers.
3. Patients free from any visible oral lesions other than the oral ulcers of BD.
4. Patient who will agree to participate in the study and take the supplied interventions.

Exclusion Criteria:

1. Patients with history of a severe or chronic medical condition including congestive heart failure, malignancy and active infection including tuberculosis, hepatitis and human immunodeficiency virus.
2. Patients who refuse to sign the informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
oral ulcer severity | During the first week (days 1, 3, and 7), then every week for 3 weeks, afterward every month for 2 months.
  oral ulcer severity score (OUSS). OUSS indicates the disease activity in recurrent oral ulcers., as the change in the numerical score reflects the change in ulcer severity in response to treatment

SECONDARY OUTCOMES:
Pain associated with oral ulcers | During the first week (days 1, 3, and 7), then every week for 3 weeks, afterward every month for 2 months.
  pain from oral ulcers will be assessed through visual analogue scale
Number of oral ulcers | During the first week (days 1, 3, and 7), then every week for 3 weeks, afterward every month for 2 months.
  Number of oral ulcers will be determined through clinical examination
healing time of oral ulcers | During the first week (days 1, 3, and 7), then every week for 3 weeks, afterward every month for 2 months.
  healing time of oral ulcers will be determined through clinical examination

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akagi S, Fujiwara T, Nishida M, Okuda A, Nagao Y, Okuda T, Tokuda H, Takayanagi K. The effectiveness of rebamipide mouthwash therapy for radiotherapy and chemoradiotherapy-induced oral mucositis in patients with head and neck cancer: a systematic review and meta-analysis. J Pharm Health Care Sci. 2019 Jul 25;5:16. doi: 10.1186/s40780-019-0146-2. eCollection 2019. PMID 31367460
- [Background] Alibaz-Oner F, Direskeneli H. Advances in the Treatment of Behcet's Disease. Curr Rheumatol Rep. 2021 May 20;23(6):47. doi: 10.1007/s11926-021-01011-z. PMID 34014377
- [Background] Ghate JV, Jorizzo JL. Behcet's disease and complex aphthosis. J Am Acad Dermatol. 1999 Jan;40(1):1-18; quiz 19-20. doi: 10.1016/s0190-9622(99)70523-2. PMID 9922007
- [Background] Hatemi G, Melikoglu M, Tunc R, Korkmaz C, Turgut Ozturk B, Mat C, Merkel PA, Calamia KT, Liu Z, Pineda L, Stevens RM, Yazici H, Yazici Y. Apremilast for Behcet's syndrome--a phase 2, placebo-controlled study. N Engl J Med. 2015 Apr 16;372(16):1510-8. doi: 10.1056/NEJMoa1408684. PMID 25875256
- [Background] Hatemi G, Merkel PA, Hamuryudan V, Boers M, Direskeneli H, Aydin SZ, Yazici H. Outcome measures used in clinical trials for Behcet syndrome: a systematic review. J Rheumatol. 2014 Mar;41(3):599-612. doi: 10.3899/jrheum.131249. Epub 2014 Feb 1. PMID 24488418
- [Background] International Team for the Revision of the International Criteria for Behcet's Disease (ITR-ICBD). The International Criteria for Behcet's Disease (ICBD): a collaborative study of 27 countries on the sensitivity and specificity of the new criteria. J Eur Acad Dermatol Venereol. 2014 Mar;28(3):338-47. doi: 10.1111/jdv.12107. Epub 2013 Feb 26. PMID 23441863
- [Background] Kudur MH, Hulmani M. Rebamipide: A Novel Agent in the Treatment of Recurrent Aphthous Ulcer and Behcet's Syndrome. Indian J Dermatol. 2013 Sep;58(5):352-4. doi: 10.4103/0019-5154.117298. PMID 24082178
- [Background] Leccese P, Ozguler Y, Christensen R, Esatoglu SN, Bang D, Bodaghi B, Celik AF, Fortune F, Gaudric J, Gul A, Kotter I, Mahr A, Moots RJ, Richter J, Saadoun D, Salvarani C, Scuderi F, Sfikakis PP, Siva A, Stanford M, Tugal-Tutkun I, West R, Yurdakul S, Olivieri I, Yazici H, Hatemi G. Management of skin, mucosa and joint involvement of Behcet's syndrome: A systematic review for update of the EULAR recommendations for the management of Behcet's syndrome. Semin Arthritis Rheum. 2019 Feb;48(4):752-762. doi: 10.1016/j.semarthrit.2018.05.008. Epub 2018 May 19. PMID 29954598
- [Background] Matsuda T, Ohno S, Hirohata S, Miyanaga Y, Ujihara H, Inaba G, Nakamura S, Tanaka S, Kogure M, Mizushima Y. Efficacy of rebamipide as adjunctive therapy in the treatment of recurrent oral aphthous ulcers in patients with Behcet's disease: a randomised, double-blind, placebo-controlled study. Drugs R D. 2003;4(1):19-28. doi: 10.2165/00126839-200304010-00002. PMID 12568631
- [Background] Nagai N, Seiriki R, Deguchi S, Otake H, Hiramatsu N, Sasaki H, Yamamoto N. Hydrogel Formulations Incorporating Drug Nanocrystals Enhance the Therapeutic Effect of Rebamipide in a Hamster Model for Oral Mucositis. Pharmaceutics. 2020 Jun 9;12(6):532. doi: 10.3390/pharmaceutics12060532. PMID 32527029
- [Background] Novak T, Hamedi M, Bergmeier LA, Fortune F, Hagi-Pavli E. Saliva and Serum Cytokine Profiles During Oral Ulceration in Behcet's Disease. Front Immunol. 2021 Dec 22;12:724900. doi: 10.3389/fimmu.2021.724900. eCollection 2021. PMID 35003055
- [Background] Quijano D, Rodriguez M. [Topical corticosteroids in recurrent aphthous stomatitis. Systematic review]. Acta Otorrinolaringol Esp. 2008 Jun-Jul;59(6):298-307. Spanish. PMID 18588791
- [Background] Senusi A, Kang A, Buchanan JAG, Adesanya A, Aloraini G, Stanford M, Fortune F. New mouthwash: an efficacious intervention for oral ulceration associated with Behcet's disease. Br J Oral Maxillofac Surg. 2020 Oct;58(8):1034-1039. doi: 10.1016/j.bjoms.2020.07.027. Epub 2020 Jul 25. PMID 32819746
- [Background] Tappuni AR, Kovacevic T, Shirlaw PJ, Challacombe SJ. Clinical assessment of disease severity in recurrent aphthous stomatitis. J Oral Pathol Med. 2013 Sep;42(8):635-41. doi: 10.1111/jop.12059. Epub 2013 Mar 19. PMID 23509958
- [Background] Taylor J, Glenny AM, Walsh T, Brocklehurst P, Riley P, Gorodkin R, Pemberton MN. Interventions for the management of oral ulcers in Behcet's disease. Cochrane Database Syst Rev. 2014 Sep 25;2014(9):CD011018. doi: 10.1002/14651858.CD011018.pub2. PMID 25254615
- [Background] Zeidan MJ, Saadoun D, Garrido M, Klatzmann D, Six A, Cacoub P. Behcet's disease physiopathology: a contemporary review. Auto Immun Highlights. 2016 Dec;7(1):4. doi: 10.1007/s13317-016-0074-1. Epub 2016 Feb 12. PMID 26868128